CLINICAL TRIAL: NCT01891539
Title: Observational Prospective Study on Chemoembolization Using Doxorubicin Drug-eluting Bead in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Observational Prospective Study on Chemoembolization With Doxorubicin for Unresectable Hepatocellular Carcinoma
Acronym: DEBDOX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Group of Endovascular Oncology (Other)
Responsible Party: Principal Investigator, Giammaria Fiorentini, Dr., International Group of Endovascular Oncology
Other Study IDs: DEBDOX01
Record Dates: First submitted 2013-06-26; First posted 2013-07-03 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Liver Cell Carcinoma Non-resectable
Keywords: Hepatocellular carcinoma, doxorubicin, chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- doxorubicin: Day +1:
  Lobar Infusion ( lobe with dominant disease) of Doxorubicin preloaded into 2 ml of drug-eluting microspheres.
  Second lobar infusion of Doxorubicin preloaded into 2 ml of drug eluting microspheres can be administered at the same time contralaterally or in a further TACE Day +30: The above procedure is repeated. Day +90: In case of response, a third administration following the above procedures will be repeated

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common type of cancer in men and the seventh in women and is the third most common cause of death from cancer worldwide. The overall incidence of HCC remains high in developing countries and is steadily rising in most industrialized countries.

TACE with Doxorubicin-eluting beads (DEB-TACE) has recently been developed as a novel therapy option for HCC. In order to maximize its therapeutic efficacy, doxorubicin-loaded beads were developed to deliver higher doses of the chemotherapeutic agent and to prolong its permanence within the tumor. The comparison of efficacy and safety of TACE with drug-eluting microspheres in comparison with conventional TACE (cTACE) showed that response and time to progression in the group was significantly higher than that of the cTACE group. TACE with drug-eluting microspheres thus appears to be a feasible and promising approach to the treatment of HCC.

This study's purpose is evaluating treatment efficacy, survival rate and safety of TACE using drug-eluting microspheres loaded with doxorubicin for unresectable hepatocellular carcinoma.

DETAILED DESCRIPTION:
This study's purpose is to assess treatment efficacy, survival rate and safety of TACE using drug-eluting microspheres loaded with doxorubicin for unresectable hepatocellular carcinoma.

Study Design: Prospective observational study . Primary objective: To collect data on tumor response after administration of drug-eluting microspheres that were preloaded with doxorubicin.

Secondary objectives: To collect data on survival rate, time to progression, tolerability of treatment, number of treatment required to achieve objective response and improvement of quality of life.

Treatment method:

Day -1 Doxorubicin at a dose of 35/50 mg/m2 has been charged onto 2 ml of microspheres at Pharmacy. It is suggested to dissolve Doxorubicin powder with 2 ml of contrast medium. The charging time of microspheres is at least 30 minutes.

Day 0: prehydration, antibiotic prophylaxis and setting up of a therapeutic scheme appropriate for analgesic prophylaxis (3-day duration) as previously reported (17)

Day +1:

Upon admittance to the radiology room, 1 vial of tropisetron (diluted in 100ml of physiological solution) and 1 vial of morphine hydrochloride diluted in 100 ml i.v. are administered by slow drip.

One vial of morphine hydrochloride diluted in 100 ml i.v. to be repeated one hour after the procedure and if necessary also after 6 hours.

Tropisetron i.v. if needed. Intra-arterial premedication (optional) with 1 vial of verapamil diluted in 4 ml of normal saline solution followed by 4 ml of lidocaine.

Tumor Infusion (segment/s with dominant disease) of Doxorubicin at a dose of 35/50 mg/m2 preloaded into 2 ml of 70-150 µm M1 microspheres.

A second tumor infusion is allowed if other lesions are present (daughter tumor), using Doxorubicin at a dose of 35/50 mg/m2 preloaded into 2 ml of 70-150 µm M1 microspheres (following radiologist and oncologist ' s planning of cure).

Day +30: The above procedure is repeated. Day +90: In case of response, a third administration following the above procedures will be repeated

Evaluation of response Response is assessed at 30, 90 and 180 days after TACE, monitoring tumor dimension using Chest-abdomen CAT scan with and without contrast medium, and cancer markers (CEA, Carbohydrate Antigen (CA) 19.9) Tumor response is performed according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria.

Assessment of quality of life Assessment of quality of life with alliative Performance Scale PPSv2 is performed during the baseline visit and 30, 60 and 180 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of HCC
2. Patient with HCC not suitable for radical therapies such as resection, liver transplantation or percutaneous therapies or patient is indicated for these therapies but there is a contraindication for them or patient rejects the above treatments
3. Multinodular or single nodular tumor more than 5cm
4. Hypervascular lesion showing contrast enhancement in the early stage after contrast media injection during CT or MRI.
5. At least one uni-dimensional lesion measurable according to the Modified RECIST criteria by CT-scan or MRI
6. No invasion in the blood vessel (hepatic portal, hepatic vein) or bile duct
7. Eastern Cooperative Oncology Group performance status is 0 - 1
8. Proper blood, liver, renal, heart functionality
9. more than 18 years old
10. Expected survival more than 6 months
11. Prior written consent

Exclusion Criteria:

1. Extrahepatic metastasis (Any lymph nodes measuring ≥ 10mm along the short axis)
2. Tumor burden involving more than 50% of the liver
3. History of biliary tract repair or endoscopic biliary tract treatment
4. Clinically important refractory ascites or pleural fluid
5. Any contraindications for hepatic embolization procedures
6. Any contraindication for doxorubicin administration
7. Contrast media allergy contraindicating angiography
8. Acute or active cardiac, hepatic or renal diseases
9. Pregnant, nursing or childbearing age women and men who are sexually active and don't want to or can't do contraception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
tumor response | 4 months
  CT scan evaluation according to RECIST 1.1

SECONDARY OUTCOMES:
survival rate | one year
  patients alive after 12 months
time to progression | 1 year
  time from start of therapy to progression

CONTACTS AND LOCATIONS:
Overall Officials: Giammaria Fiorentini, MD, Principal Investigator — International Group of Endovascular Oncology
Locations (1):
- Azienda Ospedaliera Ospedali Riuniti Marche Nord, Presidio Ospedaliero San Salvatore, Pesaro, PU, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fiorentini G. A new tool to enhance the efficacy of chemoembolization to treat primary and metastatic hepatic tumors. Expert Opin Drug Deliv. 2011 Apr;8(4):409-13. doi: 10.1517/17425247.2011.565327. Epub 2011 Mar 18. PMID 21413909
- [Result] Fiorentini G, Campanini A, Dazzi C, Davitti B, Graziani G, Priori T, Ricci Bitti R, Angelini L. Chemoembolization in liver malignant involvement. Experiences on 17 cases. Minerva Chir. 1994 Apr;49(4):281-5. PMID 8072703
- See also: International group of endovascular oncology (IGEVO) website — http://igevo.jimdo.com/